CLINICAL TRIAL: NCT05573711
Title: Determination of the Frequency of Restless Legs Syndrome and Associated Factors in People With Neuromyelitis Optica Spectrum Disorder
Brief Title: Restless Legs Syndrome in People With Neuromyelitis Optica Spectrum Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Serkan Ozakbas, MD, Dokuz Eylul University
Other Study IDs: 7304-GOA
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Neuromyelitis Optica; Restless Legs Syndrome
Keywords: sleep; neuromyelitis optica; cognitive functions
MeSH Terms: conditions — Neuromyelitis Optica; Restless Legs Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: assessments — Assessments, no specific intervention

SUMMARY:
Restless legs syndrome (RLS) is a neurological movement disorder characterized by uncomfortable and uncontrollable sensations, usually in the legs, that increase at rest, and an urge to move the legs or other affected extremities. The exact cause of RLS is unknown, but there are idiopathic and secondary forms of RLS associated with various medical conditions such as anemia, pregnancy, uremia, neuropathies, rheumatoid arthritis, parkinson's disease, spinocerebellar ataxia, and neurological disorders such as multiple sclerosis.

Neuromyelitis optica (NMO) is a severe inflammatory disease of the central nervous system.

NMO, once considered a variant of multiple sclerosis, is now recognized as a separate disease entity. In 2004, the water channel protein-specific antibody called aquaporin 4 (AQP4) was found to cause NMO, leading to the identification of NMO as a separate disease. When initially described, the disease was thought to show only necrotic and demyelinating lesions in the optic nerve and spinal cord. It was therefore thought that NMO would preferentially only attack the optic nerves and spinal cord, not the brain. However, over the years, evidence from various studies has proven that various parts of the brain are also affected during the course of the disease. In addition, some patients showing features of the disease were found to be seronegative for anti-AQP4 antibodies. These findings necessitated the need to introduce a new term "neuromyelitis optica spectrum disorders (NMOSD)" to describe all the features of the disease. Although the feeling of restlessness in the legs is frequently reported as a sensory symptom by people with NMOSD, there are limited publications to investigate the relationship between RLS and NMOSD.

The primary aim of the study is to determine the frequency and severity of RLS in people with NMOSD. The second aim of the study is to compare the presence and severity of RLS, sleep quality, daytime sleepiness level, quality of life, fatigue and Magnetic Resonance Imaging (MRI) results in people with NMOSD. The third aim of the study is to compare the cognitive functions of people with RLS positive and negative NMOSD.

People with NMOSD who came to Dokuz Eylul University Medical Faculty Hospital Neurology Department MS Polyclinic for their routine check-ups, who volunteered to participate, will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with NMOSD by a neurologist
* To be willing to participate in the study.

Exclusion Criteria:

* Diagnosed severe cognitive and/or psychiatric impairment
* Having any of the conditions known to be associated with RLS, such as anemia [hemoglobin (Hb) levels <12 mg/mL], pregnancy, uremia, neuropathies, rheumatoid arthritis, and neurological diseases other than NMOSD

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: people with neuromyelitis optica spectrum disorder
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
International Restless Legs Syndrome Study Group rating scale for restless legs syndrome | Baseline
  The International Restless Legs Syndrome Study Group rating scale for restless legs syndrome is used to assess severity of the restless legs syndrome symptoms. It consists of 10 items scored by 0 to 4. Possible scores range from 0 to 40. Higher scores indicate higher severity.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | Baseline
  Detect sleep disturbances or deficits.
Epworth Sleepiness Scale | Baseline
  The Epworth Sleepiness Scale is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. The score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the score, the higher that person's average sleep propensity in daily life, or their 'daytime sleepiness'.
Modified Fatigue Impact Scale | Baseline
  The Modified Fatigue Impact Scale provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The scale consists of 21 items with a Likert-type choose options. The total score for the scale is the sum of the scores for the 21 items. Individual subscale scores for physical, cognitive, and psychosocial functioning can also be generated by calculating the sum of specific sets of items. The total score ranges from 0 to 84. Higher score indicates higher level of fatigue.
Symbol Digit Modalities Test | Baseline
  The Symbol Digit Modalities Test is used to assess information processing speed. Using a reference key, the test taker has 90 seconds to pair specific numbers with given geometric figures in the Symbol Digit Modalities Test. The correct matches are calculated as the test score. Higher scores indicate better information processing speed.
California Verbal Learning Test-II | Baseline
  The California Verbal Learning Test-II is used to assess verbal memory. Higher scores indicate better verbal memory.
Revised Brief Visuospatial Memory Test | Baseline
  The Revised Brief Visuospatial Memory Test is used to assess visuospatial memory. Higher scores indicate better visuospatial memory.
Magnetic Resonance Imagery | Baseline
  The MRI results of the people with NMOSD included in the study, taken within the last 6 months, will be examined. Black hole, active lesion and spinal lesion presence, region and number will be noted. MRI results will be evaluated by neurologists specialized in demyelinating diseases.

OTHER OUTCOMES:
Restless Legs Syndrome Diagnostic Criteria | Baseline
  Diagnostic Criteria for Restless Legs Syndrome was developed by the Restless Legs Syndrome Working Group in 1995 and revised in 2003 and 2014. These criteria include; the need to move the legs due to uncomfortable or unpleasant sensations in the legs, the need for movement or disturbing sensations start or worsen at rest, the need for movement or disturbing sensations can be partially or totally relieved by movements such as walking or stretching, the need for movement or disturbing sensations may worsen at night or only occur in the evening or night, The aforementioned features cannot be considered only in relation to primary symptoms or other medical or behavioral conditions (e.g., myalgia, venous stasis, leg edema, leg cramps, habitual foot swing). Patients meeting all of the criteria are diagnosed with restless legs syndrome. The restless legs syndrome diagnosis will be confirmed by a neurologist.
Expanded Disability Status Scale | Baseline
  The Expanded Disability Status Scale is a method of quantifying disability in multiple sclerosis. The scale is based on a neurological examination by a clinician. It has steps from 0 to 10. The higher scores indicate higher neurological disability.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Ozakbas, MD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided